CLINICAL TRIAL: NCT03599986
Title: A Phase IV, Multi-Centric, Prospective, Observational Study to Assess the Clinical Efficacy and Safety of Leflunomide in Egyptian Patients With Active Rheumatoid Arthritis
Brief Title: Clinical Efficacy and Safety of Leflunomide in Egyptian Patients With Active Rheumatoid Arthritis
Acronym: CLEAR
Status: Completed | Type: Observational
Sponsor: Eva Pharma (Industry)
Collaborators: DataClin (Industry)
Responsible Party: Principal Investigator, Adel Mahmoud Elsayed, Professor of Internal Medicine, Rheumatology and Immunology, Eva Pharma
Other Study IDs: EVA_CLEAR_11022017
Record Dates: First submitted 2018-01-31; First posted 2018-07-26 (Actual); Results first posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Active Rheumatoid Arthritis
Keywords: RA

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Phase IV, Multi-Centric, Prospective, Observational Study to Assess the Clinical Efficacy and Safety of Leflunomide in Egyptian Patients with Active Rheumatoid Arthritis. (CLEAR)

DETAILED DESCRIPTION:
CLEAR is a phase IV, multi-centric, prospective, observational study to assess the clinical efficacy and safety of Leflunomide as first-line therapy and as add-on therapy to other DMARDs (such as Methotrexate, Hydroxychloroquine, Sulfasalazine) with or without Steroids use in Egyptian patients with Active Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Active Rheumatoid Arthritis patients selected according to the ACR/EULAR classification 2010 criteria with score ≥ 6 points.
2. Male or female patients aged 18-60 years old.
3. Leflunomide naïve patients or patients with previous Leflunomide administration (after at least 6 month wash out period from date of baseline visit) who will be prescribed Leflunomide at the sole decision of the treating physician.
4. Patients with or without another DMARDs including Methotrexate, Sulfasalazine and/or Hydroxychloroquine with or without steroids use who experienced therapy resistance, inadequate response or intolerance.
5. Patients read, understand and signed informed consent prior to inclusion.
6. Patients willing to complete and literate in the language of the available Health Assessment Questionnaire (HAQ Disability Index) either alone or with minimal assistance from caregivers and/or trained site personnel.

Exclusion Criteria:

1. Female patients who are pregnant or lactating at the time of inclusion or those who are planning for pregnancy within the coming year from the time of inclusion to the study.
2. Patients with contraindications to active constituent of Leflunomide.
3. Patients with severe concurrent infection (necessitating IV antibiotics or hospitalization).
4. Patients with history of non-treated hepatitis B &/or C infection.
5. Patients with history of severe liver disease (child C class).
6. Patients with history of severe renal insufficiency (creatinine clearance ≤30 ml/min.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients are between 18 and 60 years of age, with Active Rheumatoid Arthritis selected according to the ACR/EULAR classification criteria with score ≥ 6 points.
  Patients are Leflunomide naïve or with previous Leflunomide administration (after at least 6-month wash out period from date of baseline visit).
  Patients are with or without other DMARDs including Methotrexate, Sulfasalazine and/or Hydroxychloroquine with or without steroids use who experienced therapy resistance, inadequate response or intolerance.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2018-10-13 (Actual); Study Completion 2018-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adel Elsayed, MD, Principal Investigator — Professor, Department of Internal Medicine, Rheumatology and Immunology, Ain Shams University; Egypt
Locations (1):
- Private clinics, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Not yet

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Adult Egyptian patients with active rheumatoid arthritis, fulfilling the ACR/EULAR 2010 classification criteria, for whom leflunomide was prescribed, were included and followed up for 9 months.
Period: Overall Study
Arm/Group | Single Arm
Started | 398
Completed | 366
Not Completed | 32

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 366
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Row population (n=365) differs from the overall population (n=366) due to missing data.
  years
    number analyzed (Participants) | 365
    (all) | 44.1 [35.78 to 52.42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 309
  Male | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Patient's distribution per governorates [Count of Participants; unit: Participants]
  Alexandria | 108
  Assuit | 3
  Banha | 18
  Cairo | 98
  Ismailia | 32
  Mansoura | 15
  Menoufia | 27
  Minya | 17
  Zagazig | 48
Marital status [Count of Participants; unit: Participants]
  Single | 31
  Married | 312
  Divorced | 3
  Widow/widower | 20
Education [Count of Participants; unit: Participants]
  Illiterate | 31
  Basic/primary | 80
  Secondary | 120
  University/Higher | 135
Residence [Count of Participants; unit: Participants]
  Rural | 138
  Urban | 228
Birth Control [Count of Participants; unit: Participants]
  No | 151
  Yes | 135
  Missing | 80
Specification of birth control method used [Count of Participants; unit: Participants] — Population: The number analyzed (n=135) is that of patients who were using a birth control method during the study period.
  Participants
    Hormonal: number analyzed (Participants) | 135
    Hormonal | 43
    Intrauterine Device (IUD): number analyzed (Participants) | 135
    Intrauterine Device (IUD) | 85
    Barrier methods: number analyzed (Participants) | 135
    Barrier methods | 3
    Natural methods: number analyzed (Participants) | 135
    Natural methods | 3
    Unspecified: number analyzed (Participants) | 135
    Unspecified | 1
Patients currently taking medications for comorbidities [Count of Participants; unit: Participants]
  Yes | 101
  No | 265
Medications for reasons other than Rheumatoid Arthritis [Count of Participants; unit: Participants]
  Bisporolol | 27
  Methotrexate | 19
  Omeprazole | 17
  Hydrochlorothiazide | 16
  Diclofenac | 14
  Folic acid | 12
  Prednisolone | 11
  Metformin | 10
  Glucosamine | 9
  Pantoprazole | 9
  Piroxicam | 9
  Calcium | 8
  Enalapril maleate | 8
  Ergocalciferol | 8
  Chymotrypsin | 7
  Trypsin | 7
  Glimepiride | 6
  Magnesium | 6
  Calcium carbonate | 5
  Captopril | 5
  Diclofenac sodium | 5
  Pregabalin | 5
  Vitamin D | 5
  Atorvastatin | 4
  Chondroitin sulphate | 4
  Hydroxychloroquine sulphate | 4
  Ibuprofen | 4
  Levothyroxine | 4
  Meloxicam | 4
  Ranitidine | 4
  Silymarin | 4
  Vitamin B12 | 4
Age at first menstrual period [Median (Inter-Quartile Range); unit: years] — Population: The row population (n=244) differs from that of the overall female population (n=309) because the data of 65 female patients were missing.
  years
    number analyzed (Participants) | 244
    (all) | 13 [12 to 14]
Menstruation status [Count of Participants; unit: Participants] — Population: The eligible population for this analysis is the female population (n=309).
  Participants
    Menstruating: number analyzed (Participants) | 309
    Menstruating | 192
    Premenopausal: number analyzed (Participants) | 309
    Premenopausal | 8
    Menopausal: number analyzed (Participants) | 309
    Menopausal | 38
    Post-menopausal: number analyzed (Participants) | 309
    Post-menopausal | 70
    Missing: number analyzed (Participants) | 309
    Missing | 1
Regularity of menstrual periods if menstruating or premenopausal [Count of Participants; unit: Participants] — The regularity of menstrual periods in menstruating patients (n=192) and premenopausal patients (n=8). Population: The row population (n=200) is the sum of patients who were menstruating (n=192) and those who were premenopausal (n=8).
  Participants
    Regular: number analyzed (Participants) | 200
    Regular | 23
    Irregular: number analyzed (Participants) | 200
    Irregular | 161
    Missing: number analyzed (Participants) | 200
    Missing | 16
Duration of Rheumatoid Arthritis [Median (Inter-Quartile Range); unit: years] — Population: The row population (n=358) differs from the overall population (n=366) because the data of 8 patients is missing.
  years
    number analyzed (Participants) | 358
    (all) | 2.03 [-0.72 to 4.78]
Did the patient receive leflunomide before? [Count of Participants; unit: Participants]
  Yes | 51
  No | 315
Did the patient take a loading dose of leflunomide before? [Count of Participants; unit: Participants] — Population: The row population (n=51) differs from the overall population (n=366) because the analysis is concerned with patients who have previously received leflunomide during their past treatment of rheumatoid arthritis.
  Participants
    Yes: number analyzed (Participants) | 51
    Yes | 31
    No: number analyzed (Participants) | 51
    No | 20
Duration of RA treatment with medications other than leflunomide [Median (Inter-Quartile Range); unit: months] — Duration of treatment of rheumatoid arthritis (RA) with medications other than leflunomide until the time of the first study visit.
  months | 27.7 [1.63 to 53.78]
AEs/SAEs during previous treatment of RA [Count of Participants; unit: Participants]
  Yes | 94
  No | 252
  Missing | 20
X-ray performed for both hands? [Count of Participants; unit: Participants]
  Yes | 144
  No | 198
  Missing | 24
Poor prognostic factors [Count of Participants; unit: Participants] — High disease activity was determined as a measure of composite indices (DAS28, SDAI and/or CDAI).
  Participants
    Bony erosions by radiograph | 90
    High swollen joint count | 136
    Extra-articular disease | 19
    Functional limitation (HAQ) | 240
    High disease activity | 295
    High CRP and ESR or high RF and/or anti-CCP | 237
Weight [Mean (Standard Deviation); unit: Kilogram (Kg)] — Population: The row population (n=348) is different from the overall population (n=366) given that data on weight is missing from 18 patients.
  Kilogram (Kg)
    number analyzed (Participants) | 348
    (all) | 81.3 (15.25)
Height [Mean (Standard Deviation); unit: Centimeter (cm)] — Population: The number analyzed in row (n=346) differs from the overall population (n=366) because height data is missing from 20 patients.
  Centimeter (cm)
    number analyzed (Participants) | 346
    (all) | 164 (12.19)
Heart rate [Mean (Standard Deviation); unit: beats/minute] — Population: The row population (n=364) differs from the overall population (n=366) because data on heart rate was missing from 2 patients.
  beats/minute
    number analyzed (Participants) | 364
    (all) | 81.7 (8.3)
Temperature [Mean (Standard Deviation); unit: Degrees Celsius] — Population: The row population (n=359) differs from that of the overall population (n=366) because the temperature data of 7 patients were missing.
  Degrees Celsius
    number analyzed (Participants) | 359
    (all) | 37.2 (2.7)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 121.9 (13.66)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Data on diastolic blood pressure is missing from 1 patient.
  mmHg
    number analyzed (Participants) | 365
    (all) | 78.36 (7.89)
Physical Examination outcome [Count of Participants; unit: Participants] — Population: The row population (n=359) differs from the overall population (n=366) because data on physical examination outcome is missing from 7 patients.
  Participants
    Normal: number analyzed (Participants) | 359
    Normal | 312
    Abnormal: number analyzed (Participants) | 359
    Abnormal | 47
Smoking status [Count of Participants; unit: Participants] — Population: The row population (n=364) is different than that of the overall population (n=366) because data on the smoking status of 2 patients is missing.
  Participants
    Never: number analyzed (Participants) | 364
    Never | 333
    Former: number analyzed (Participants) | 364
    Former | 9
    Current: number analyzed (Participants) | 364
    Current | 22
Status of alcohol consumption [Count of Participants; unit: Participants] — Population: The row population (n=363) differs from the overall population (n=366) because data on the status of alcohol consumption is missing from 3 patients.
  Participants
    Never: number analyzed (Participants) | 363
    Never | 363
    Yes: number analyzed (Participants) | 363
    Yes | 0
    Missing | 3
Patients with comorbidities [Count of Participants; unit: Participants]
  Yes | 115
  No | 251
Comorbidities [Count of Participants; unit: Participants]
  Hypertension | 60
  Atherosclerosis | 1
  Coronary artery disease | 3
  Myocardial infarction | 1
  Stroke | 1
  Peripheral Vascular Disease | 1
  Diabetes Mellitus II | 21
  Obesity | 32
  Dyslipidemia | 10
  Respiratory and thoracic disorders | 6
  GIT disorders | 10
  Hepatobiliary disorders | 1
  Nervous system disorders | 5
  Psychiatric disorders | 1
  Reproductive system disorders | 2
  Musculoskeletal disoders | 28
  Autoimmune disease | 10
  Other | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Remission, Low, Moderate or High Disease Activity (in Terms of CDAI Scores) in Visits 1 and 6.
Description: Assessing the clinical efficacy of leflunomide as first-line therapy and as add-on therapy to other DMARDs, with or without steroids in Egyptian patients with active rheumatoid arthritis [in terms of the number of patients in remission (i.e. CDAI score 0.0 - 2.8), of low disease activity (i.e. CDAI score 2.9 - 10.0), of moderate disease activity (i.e. CDAI score 10.1 - 22.0) and of high disease activity (i.e. CDAI score 22.1 - 76.0) in visits 1 (at baseline) and 6 (at week 36)].
  CDAI score: The sum of Tender joint score, Swollen joint score, Patient global score, and Patient global score.
  CDAI score interpretation:
  0.0 - 2.8: Remission 2.9 - 10.0: Low Activity 10.1 - 22.0: Moderate Activity 22.1 - 76.0: High Activity
Time Frame: 9 months
Population: Only patients with at least one treatment dose and post-assessment score of last observation carried forward (LOCF) convention were analyzed in terms of efficacy endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 366
Participants
  Disease Severity: Remission : Visit 1 | 0
  Disease Severity: Remission : Visit 6 | 70
  Disease severity: Low activity : Visit 1 | 10
  Disease severity: Low activity : Visit 6 | 116
  Disease severity: Moderate activity : Visit 1 | 53
  Disease severity: Moderate activity : Visit 6 | 113
  Disease severity: High activity : Visit 1 | 303
  Disease severity: High activity : Visit 6 | 67

2. Primary Outcome: Number of Patients With Different Disability Scores in Terms of the Mean Relative Change in Health Assessment Questionnaire - Disability Index Score on Visits 1 and 6.
Description: Assessing the clinical efficacy of leflunomide as first-line therapy and as add-on therapy to other DMARDs, with or without steroids in Egyptian patients with active rheumatoid arthritis [in terms of the number of patients with mild difficulties to moderate disability, moderate to severe disability and severe to very severe disability; according to the mean relative change in health assessment questionnaire - disability index score (HAQ-DI) at visits 1 (at baseline) and 6 (at week 36)].
  A HAQ-DI score of 0.0 - 1 indicates mild difficulties to moderate disability, a HAQ-DI score of 1.1 - 2 indicates moderate to severe disability and a HAQ-DI score of 2.1 - 3 indicates severe to very severe disability.
  There are eight categories; first score within each category: Dressing and Grooming, Arising, Eating, Walking, Hygiene, Reach, Grip, and Activities.
  Total score is the mean of the eight category scores. Higher scores indicate greater disability.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm: Adult Egyptian patients with active rheumatoid arthritis, fulfilling the ACR/EULAR 2010 classification criteria, for whom leflunomide was prescribed for 9 months.
Arm/Group | Single Arm
Number analyzed (Participants) | 366
Participants
  HAQ score 0.0 - 1 : Visit 1 | 112
  HAQ score 0.0 - 1 : Visit 6 | 318
  HAQ score 1.1 - 2 : Visit 1 | 200
  HAQ score 1.1 - 2 : Visit 6 | 43
  HAQ score 2.1 - 3 : Visit 1 | 54
  HAQ score 2.1 - 3 : Visit 6 | 5

3. Secondary Outcome: Number of Adverse Events (AEs)/ Serious Adverse Events (SAEs) Experienced by Rheumatoid Arthritis Patients Receiving Leflunomide as First-line Therapy and as add-on Therapy to Other DMARD, With or Without Steroids and Their Relation to Study Medication.
Description: Identifying the safety profile of leflunomide whether used as first-line therapy and/or as add-on therapy to other DMARDs with or without steroids in Egyptian patients with active rheumatoid arthritis.
Time Frame: 9 months
Population: In the safety population (n = 398), 23 adverse events were experienced. These are listed in the table.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 398
Participants
  Hepatic enzyme increased | 6
  Swollen/tender joint count increased | 2
  White blood cell count decreased | 2
  Abdominal discomfort | 2
  Cardiac death | 1
  Anemia | 1
  Bicytopenia | 1
  Flushing/hyperhidrosis/dry mouth/lip disoloration | 1
  Hypertension | 1
  Oropharyngeal pain | 1
  Purpura | 1
  Rheumatoid arthritis | 1
  Scleritis | 1
  Supraventricular tachycardia | 1
  Diarrhea | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between visit 2 (at week 6) and visit 6 (at week 36); making the time frame of collecting safety data 30 weeks.
Description: An adverse event was defined as any untoward medical occurrence in a clinical investigation subject associated with the use of a product or a medical device; the event does not necessarily need to have a causal relationship with the treatment or usage. A serious adverse event was defined as that from clinicaltrials.gov.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/398
Serious Adverse Events (participants affected / at risk) | 0/398
Other Adverse Events (participants affected / at risk) | 20/398
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=398)
Hepatic Enzyme increase (Hepatobiliary disorders) | 6
Swollen/Tender joint count increased (Musculoskeletal and connective tissue disorders) | 2
White blood cell count decreased (Blood and lymphatic system disorders) | 2
Abdominal discomfort (General disorders) | 2
Cardiac death (Cardiac disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Bicytopenia (Blood and lymphatic system disorders) | 1
Flushing/hyperhidrosis/dry mouth/lip discoloration (General disorders) | 1
Hypertension (Cardiac disorders) | 1
Oropharyngeal pain (General disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rheumatoid Arthritis (Immune system disorders) | 1
Scleritis (Eye disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03599986/Prot_SAP_000.pdf